CLINICAL TRIAL: NCT02265250
Title: Pilot Study-Magnetic Resonance Imaging for Global Atherosclerosis Risk Assessment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Janet Wei, Co-Principal Investigator, Cedars-Sinai Medical Center
Other Study IDs: Pro00037025
Record Dates: First submitted 2014-10-03; First posted 2014-10-15 (Estimated); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: Cardiovascular Disease; Atherosclerosis
Keywords: magnetic resonance imaging; positron emission tomography
MeSH Terms: conditions — Cardiovascular Diseases; Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — We will obtain fasting lipid and inflammatory biomarkers (LDL-C, HDL-C, lipoprotein(a), ApoB/ApoA-1 ratio, hemoglobin A1c, plasma adiponectin, hsCRP).
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Asymptomatic, CACS <300: 5 asymptomatic subjects with low CVD risk, defined as recent coronary artery calcium score (CACS) <300
  Noncontrast MRI of the bilateral carotid, coronary, and superficial femoral arteries; Laboratory blood test (cardiovascular biomarkers)
  Interventions: Other: MRI; Other: Laboratory blood test
- Asymptomatic, CACS ≥300: 5 asymptomatic subjects with increased CVD risk, defined as a recent coronary artery calcium score (CACS) ≥300
  Noncontrast MRI of the bilateral carotid, coronary, and superficial femoral arteries; Laboratory blood test (cardiovascular biomarkers); Simultaneous 18F-NaF PET/MRI of the bilateral carotid, coronary, and superficial femoral arteries
  Interventions: Other: MRI; Other: PET/MRI; Other: Laboratory blood test
- Stable angina: 5 subjects with stable angina and evidence of coronary atherosclerosis based on a recent invasive or CT coronary angiogram
  Noncontrast MRI of the bilateral carotid, coronary, and superficial femoral arteries; Laboratory blood test (cardiovascular biomarkers); Simultaneous 18F-NaF PET/MRI of the bilateral carotid, coronary, and superficial femoral arteries
  Interventions: Other: MRI; Other: PET/MRI; Other: Laboratory blood test
- Recent acute MI: 5 subjects with a recent acute myocardial infarction (within 1 month) and evidence of coronary atherosclerosis based on invasive or CT coronary angiogram
  Noncontrast MRI of the bilateral carotid, coronary, and superficial femoral arteries; Laboratory blood test (cardiovascular biomarkers); Simultaneous 18F-NaF PET/MRI of the bilateral carotid, coronary, and superficial femoral arteries
  Interventions: Other: MRI; Other: PET/MRI; Other: Laboratory blood test

INTERVENTIONS:
Other: MRI — Noncontrast T1- and T2-weighted 3.0 T MRI of the bilateral carotid, coronary, and superficial femoral arteries
Other: PET/MRI — Simultaneous 18F-NaF PET/MRI of the bilateral carotid, coronary, and superficial femoral arteries
  Groups: Asymptomatic, CACS ≥300; Recent acute MI; Stable angina
Other: Laboratory blood test — Cardiovascular biomarkers

SUMMARY:
Cardiovascular disease (CVD) remains the leading cause of death in the United States, and improved CVD risk assessment is needed for personalized medicine. Atherosclerosis measures including plaque volume and adverse plaque features have prognostic value. Novel techniques have been developed for assessing carotid, coronary, and femoral atherosclerosis using magnetic resonance imaging (MRI) methods that are rapid and reproducible, have improved spatial resolution, and do not require contrast media, making atherosclerosis assessment in multiple vascular beds feasible during a single MRI session. This pilot research will provide preliminary data to develop an innovative global atherosclerosis measure including carotid, coronary, and femoral vascular beds, for assessing cardiovascular risk and for monitoring atherosclerosis response to therapy. 20 participants will be recruited in one year.

DETAILED DESCRIPTION:
There are up to 2 study visits in this study.

During the first visit, the investigators will obtain non-contrast MRI (carotid, coronary, and femoral) in 20 subjects with known coronary atherosclerosis but varying degrees of CVD risk.

1. 5 asymptomatic subjects with lower CVD risk (recent coronary artery calcium score [CACS] 10-299)
2. 5 asymptomatic subjects with higher CVD risk (CACS 300-1000)
3. 5 subjects with known coronary atherosclerosis and stable angina
4. 5 subjects with known atherosclerosis and recent acute myocardial infarction

The investigators will measure plaque volume and assess adverse plaque features (intra-plaque hemorrhage, positive remodeling, lesion eccentricity) in the three vascular beds.

Eight of these subjects with evidence of large plaque burden by MRI will be asked to return for a simultaneous positron emission tomography (PET)-MRI imaging with 18F-sodium fluoride (18F-NaF) of their carotid, coronary, and femoral arteries, in which 18F-NaF uptake in plaque will represent micro-calcifications, which is associated with high-risk plaque.

In all 20 subjects, the investigators will also measure the following biomarkers which have been shown to be useful for CVD risk assessment of atherosclerosis: LDL, HDL, lipoprotein(a), apolipoprotein B/A-1 ratio, hemoglobin A1c, adiponectin, and highly sensitive C-reactive protein. The investigators will also calculate their estimated 10-year and lifetime atherosclerotic CVD risk (American Heart Association), Framingham 10-year CVD risk, and Reynolds 10-year CVD risk scores.

We aim to obtain the second scan within 3 months of the first visit; thus, the subjects will participate in the study for approximately 3 months.

All the procedures are research-related. The research visit will take approximately 3 hours, and there will be maximum two visits. There are no collaborations with other sites.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women with evidence of coronary atherosclerosis based on a recent CACS 10-1000 or an invasive or CT coronary angiogram (within 6 weeks of recruitment)
2. No planned revascularization procedures

Exclusion Criteria:

1. Contraindications to MRI
2. Pregnant and lactating women
3. Body mass index (BMI)>40
4. Active smoking
5. Resting heart rate>75 beats per minute
6. Arrhythmia
7. Prior carotid/coronary/peripheral revascularization
8. Life expectancy <5 years
9. Allergy to animal dander
10. Severe asthma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 20 subjects with known coronary atherosclerosis but varying degrees of CVD risk
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2014-09; Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Plaque Volume | 24 hours
  Quantitative plaque measurement using MRI software (VesselMass)
Adverse plaque features | 24 hours
  Presence of positive remodeling, lesion eccentricity, and intraplaque hemorrhage of plaque, on MRI

SECONDARY OUTCOMES:
18F-NaF PET uptake | 3-6 months
  Measured as maximum tissue/background ratio (TBR), to assess for high-risk plaque
Laboratory biomarkers | 24 hours
  Measured as levels of LDL-C, HDL-C, lipoprotein(a), ApoB/ApoA-1 ratio, hemoglobin A1c, plasma adiponectin, hsCRP
Clinical risk scores | 24 hours
  Measured as (1) ACC/AHA 10-year and lifetime atherosclerotic CVD risk, (2) Framingham 10-year CVD risk, and (3) Reynolds Risk 10-year CVD risk

CONTACTS AND LOCATIONS:
Overall Officials: Janet Wei, MD, Principal Investigator — Cedars-Sinai Medical Center; Noel Bairey Merz, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes